CLINICAL TRIAL: NCT01706718
Title: The Effects of Beetroot Enriched Bread on Postprandial Vascular Function, Arterial Stiffness and Blood Pressure in Healthy Men
Brief Title: Beetroot Enriched Bread, Blood Pressure and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 10/18; University of Reading (Other: University of Reading)
Record Dates: First submitted 2012-09-27; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Hypertension
Keywords: Beetroot; Blood pressure; Vascular function
MeSH Terms: conditions — Hypertension | interventions — Bread

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control white bread (Placebo Comparator)
  Interventions: Dietary Supplement: Bread
- Beetroot bread (Experimental)
  Interventions: Dietary Supplement: Bread

INTERVENTIONS:
Dietary Supplement: Bread

SUMMARY:
Dietary nitrate is known to lower blood pressure. Beetroot is a rich source of nitrate and could therefore be an important dietary component in the management of hypertension and cardiovascular disease, however consumption is relatively low. We evaluated the effects of beetroot enriched bread ingestion on acute microvascular reactivity, arterial stiffness and blood pressure response in healthy men.

ELIGIBILITY:
Inclusion Criteria:

* Male
* A signed consent form
* Age 18-64 years
* Body mass index - 18.5-30 kg/m2
* Non-smoking, healthy individuals
* Normal blood pressure at screening (< 150/90)

Exclusion Criteria:

* Subjects with anaemia
* Sufferers of chronic illnesses
* Individuals with food allergies
* People with diabetes
* People with coeliac disease
* Women
* Vegetarians

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Vascular reactivity | Change from baseline at 2, 4 and 6 hours after bread consumption
  Forearm blood flow by Laser Doppler Imaging with iontophoresis

SECONDARY OUTCOMES:
Arterial stiffness | Change from baseline at 2, 4 and 6 hours after bread consumption
  Pulse wave analysis (PWA) and velocity (PWV)
Blood pressure | Change from baseline at 30 minute intervals for 7 hours
  By ambulatory blood pressure monitor
Plasma nitrate | Every 30 minutes for 7 hours
Plasma nitrite | Every 30 minutes for 7 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Background] Hobbs DA, Kaffa N, George TW, Methven L, Lovegrove JA. Blood pressure-lowering effects of beetroot juice and novel beetroot-enriched bread products in normotensive male subjects. Br J Nutr. 2012 Dec 14;108(11):2066-74. doi: 10.1017/S0007114512000190. Epub 2012 Mar 14. PMID 22414688
- [Derived] Hobbs DA, Goulding MG, Nguyen A, Malaver T, Walker CF, George TW, Methven L, Lovegrove JA. Acute ingestion of beetroot bread increases endothelium-independent vasodilation and lowers diastolic blood pressure in healthy men: a randomized controlled trial. J Nutr. 2013 Sep;143(9):1399-405. doi: 10.3945/jn.113.175778. Epub 2013 Jul 24. PMID 23884387